CLINICAL TRIAL: NCT01694563
Title: AtriCure Synergy Ablation Lesions for Non-Paroxysmal Forms of Atrial Fibrillation Treatment During Concomitant On-Pump Endo/Epicardial Cardiac Surgery
Brief Title: ABLATE Post Approval Study - Synergy Ablation Lesions for Non-Paroxysmal Atrial Fibrillation
Acronym: ABLATE-PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2011-1; NCT01174745 (obsolete NCT alias)
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2018-03

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atrial Fibrillation (Other): Patients with non-paroxysmal atrial fibrillation (persistent or longstanding persistent)who are scheduled to undergo elective concomitant open, on-pump cardiac surgical procedure and the Maze IV ablation procedure. This single arm registry is designed to monitor the AtriCure Synergy Ablation System for continued safety and efficacy during the peri-procedural and long term phase during commercial use.
  Interventions: Device: Synergy Ablation System

INTERVENTIONS:
Device: Synergy Ablation System — Patient will undergo an elective open cardiac surgical procedure to be performed on cardiopulmonary bypass for one or more of the following:
  * Coronary Artery Bypass Grafting (CABG)
  * Mitral valve repair or replacement
  * Aortic valve repair or replacement
  * Tricuspid valve repair or replacement The aim of the treatment is a complete bi-atrial Maze IV procedure which includes pulmonary vein isolation coupled with lesions made on both the left and right atria.
  Other Names: Isolator Synergy Handpieces; Isolator Synergy Clamp

SUMMARY:
The primary objective of this post-approval study is to evaluate the clinical outcomes in a cohort of patients with non-paroxysmal forms of atrial fibrillation (persistent or long-standing persistent) treated during commercial use of the AtriCure Synergy Ablation System by physicians performed the Maze IV procedure.

DETAILED DESCRIPTION:
This prospective, open label, multi-center, observational, single arm registry is designed to monitor the AtriCure Synergy Ablation System continued safety and efficacy during the peri-procedural and long-term phase during commercial use in patients being treated for non-paroxysmal forms of atrial fibrillation who are undergoing a concomitant open, on-pump cardiac surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years of age
* History of non-paroxysmal form of Atrial Fibrillation (AF) as defined by the Heart Rhythm Society/European Heart Rhythm Association/European Cardiac Arrhythmia Society Consensus Statement:

  * Persistent AF shall be defined as continuous AF that is sustained beyond seven days. Episodes of AF in which a decision is made to electrically or pharmacologically cardiovert the patient after greater than or equal to 48 hours of AF but prior to 7 days, should also be classified as persistent AF episodes.
  * Longstanding persistent AF shall be defined as continuous AF of greater than 12 months duration. The performance of a successful cardioversion (sinus rhythm >30 seconds) within 12 months of an ablation procedure with documented early recurrence of AF with 30 days should not alter the classification of AF as longstanding persistent.
* Subject is scheduled to undergo elective open cardiac surgical procedure(s) to be performed on cardiopulmonary bypass for one or more of the following: Coronary Artery Bypass Grafting, Mitral valve repair or replacement, Aortic valve repair or replacement, Tricuspid valve repair or replacement. In conjunction with these procedure patent foramen ovale (PFO) or atrial septal defect (ASD) repair are allowed.
* The patient (or their legally authorized representative) agrees to participate in this study by singing the Institutional Review Board (IRB) approved informed consent form.
* Willing and able to return for scheduled follow up visits.

Exclusion Criteria:

* Stand along AF without indication(s) for concomitant cardiac surgery.
* Need for emergent cardiac surgery (i.e., cardiogenic shock).
* Preoperative need for an intra-aortic balloon pump or intravenous inotropes.
* Pregnancy or desire to get pregnant for the duration of the study concomitant surgical procedure through the thirty six (36) month follow up period).
* Enrolled in another clinical trial that could confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCarthy, MD, Study Chair — Chief, Division of Cardiac Surgery, Northwestern University
Locations (49):
- United States (49):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Scottsdale Healthcare Clinical Research Institute, Scottsdale, Arizona
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Cedars-Sinai Medical Center, West Hollywood, California
  - Hartford Hospital, Hartford, Connecticut
  - Lee Memorial Hospital, Fort Myers, Florida
  - University of Florida Cardiothoracic Surgery, Gainesville, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Northside Hospital, St. Petersburg, Florida
  - James A. Haley Veteran's Hospital/Cardiothoracic Surgery, Tampa, Florida
  - Pepin Heart Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Evanston, Illinois
  - SIU- Memorial Medical Center, Springfield, Illinois
  - St. Francis Heart Hospital, Indianapolis, Indiana
  - Inidiana Heart Center, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Veteran Affairs Boston Healthcare System, West Roxbury, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - United Heart & Vascular/Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Nebraska Heart, Lincoln, Nebraska
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Mission Hospital/Asheville Heart, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Triad Cardiac and Thoracic Surgeons/Cone Health, Greensboro, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania (HUP), Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - UT Southwestern University Hospital, Dallas, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aspirus Wausau Hospital, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from: September 2012 thru October 2017
Groups:
- Atrial Fibrillation: Subjects enrolled exhibited the following types of Atrial fibrillation: Non-Paroxysmal, Persistent, and Long-Standing Persistent
Period: Overall Study
Arm/Group | Atrial Fibrillation
Started | 365
Completed | 278
Not Completed | 87

BASELINE CHARACTERISTICS:
Groups:
- Atrial Fibrillation: Patients with non-paroxysmal atrial fibrillation (persistent or longstanding persistent)who are scheduled to undergo elective concomitant open, on-pump cardiac surgical procedure and the Maze IV ablation procedure. This single arm registry is designed to monitor the AtriCure Synergy Ablation System for continued safety and efficacy during the peri-procedural and long term phase during commercial use.
  Synergy Ablation System: Patient will undergo an elective open cardiac surgical procedure to be performed on cardiopulmonary bypass for one or more of the following:
  * Coronary Artery Bypass Grafting (CABG)
  * Mitral valve repair or replacement
  * Aortic valve repair or replacement
  * Tricuspid valve repair or replacement The aim of the treatment is a complete bi-atrial Maze IV procedure which includes pulmonary vein isolation coupled with lesions made on both the left and right atria.
Arm/Group | Atrial Fibrillation
Number analyzed (Participants) | 365
Age, Continuous [Mean (Full Range); unit: years] | 69.8 [36.7 to 87.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 331
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 365
History of Arrhythmia [Count of Participants; unit: Participants] | 365

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Free From Atrial Fibrillation (AF), Atrial Flutter or Atrial Tachycardia While Off Class I and Class III Antiarrhythmic Drugs for at Least 4 Weeks.
Description: The number of participants free from atrial fibrillation (AF), i.e., episodes lasting >30 continuous seconds duration of either AF, atrial flutter or atrial tachycardia while off Class I and III antiarrythmic drugs for at least 4 weeks as determined by core last assessment of a 48 hour Holter, Zio Patch or Pacemaker Implantation (PPM) interrogation recording performed at a minimum of 36 months postoperatively.
Time Frame: 36 months post-operatively
Population: Freedom from AF and off antiarrhythmic drugs (AADs) at specific time points. The participants that met the endpoint are reflected in the Outcome Measure Data Table.
Measure: Count of Participants; unit: Participants
Groups:
- 36 Months Post-operatively: The primary effectiveness outcome is defined as the proportion of patients free from AF (i.e. no episodes lasting > 30 continuous seconds duration of either Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia) while off Class I and III antiarrhythmic drugs for at least 4 weeks as determined by an independent core lab assessment of 48 hour Holter, Zio™ Patch or PPM interrogation recording performed at a minimum of 36 months postoperatively.
Arm/Group | 36 Months Post-operatively
Number analyzed (Participants) | 232
Participants | 146
Statistical Analysis 1: Comparison: 36 Months Post-operatively; The primary effectiveness hypothesis for this study was to demonstrate a superiority success rate at 36-months follow-up in patients treated with the AtriCure Synergy Ablation System compared to a pre-established performance goal; Test type: Superiority; p = 0.05, Fisher Exact

2. Secondary Outcome: Secondary Efficacy Outcome
Description: The proportion of patients free from AF, regardless of AAD usage (i.e. no episodes lasting > 30 continuous seconds duration of either Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia), as determined by an independent core lab assessment of 48-hour Holter, Zio™ Patch or PPM interrogation recording performed at a minimum of 12,24, and 36 months post-operatively.
Time Frame: 12, 24, and 36 months post-operatively
Population: Secondary success was defined as freedom from AF regardless of antiarrhythmic drug usage. The participants that met the endpoint are reflected in the Outcome Measure Data Table.
Measure: Count of Participants; unit: Participants
Groups:
- 12 Months Post-operatively; 24 Months Post-operatively; 36 Months Post-operatively: Secondary success was defined as freedom from AF regardless of antiarrhythmic drug usage.
Arm/Group | 12 Months Post-operatively | 24 Months Post-operatively | 36 Months Post-operatively
Number analyzed (Participants) | 271 | 242 | 228
Participants | 216 | 187 | 168
Statistical Analysis 1: Comparison: 12 Months Post-operatively; Secondary success was defined as freedom from AF regardless of antiarrhythmic drug usage at 12 months post-operatively; Test type: Superiority; Clopper-Pearson = 90 — 90% confidence interval calculated using the Clopper-Pearson method
Statistical Analysis 2: Comparison: 24 Months Post-operatively; Secondary success was defined as freedom from AF regardless of antiarrhythmic drug usage at 24 months post-operatively; Test type: Superiority; Clopper-Pearson = 90 — 90% confidence interval calculated using the Clopper-Pearson method
Statistical Analysis 3: Comparison: 36 Months Post-operatively; Secondary success was defined as freedom from AF regardless of antiarrhythmic drug usage at 36 months post-operatively; Test type: Superiority; Clopper-Pearson = 90; 90% confidence interval using the Clopper-Pearson method

ADVERSE EVENTS:
Time Frame: All adverse events were collected for 36 months.
Description: An adverse event is any untoward medical occurrence (signs, symptoms, abnormal laboratory findings) in a patient regardless of relationship to the device or procedure. Each adverse event is considered to be either anticipated or unanticipated as described below. The site is required to report all adverse events that occur in the study.
Groups:
- Treatment Arm: Patients with non-paroxysmal atrial fibrillation ………..
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 20/365
Serious Adverse Events (participants affected / at risk) | 289/365
Other Adverse Events (participants affected / at risk) | 271/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=365)
Bradycardia (Cardiac disorders) | 20 (20)
Ventricular Tachycardia (Cardiac disorders) | 9 (9)
Venous Injury (Cardiac disorders) | 1 (1)
Haemorrhage (Cardiac disorders) | 1 (1)
Death (General disorders) | 20 (20)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 16 (16)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic Valve Incompetence (Cardiac disorders) | 5 (5)
Arrythmia (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 45 (45)
Atrial Flutter (Cardiac disorders) | 17 (17)
Atrial Rupture (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 2 (2)
Atrioventricular Block (Cardiac disorders) | 24 (24)
Cardiac Arrest (Cardiac disorders) | 6 (6)
Cardiac Failure (Cardiac disorders) | 90 (90)
Cardiac Tamponade (Cardiac disorders) | 5 (5)
Cardiogenic Shock (Cardiac disorders) | 14 (14)
Cardiorenal Syndrome (Cardiac disorders) | 1 (1)
Cardio-respiratory Arrest (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Complete Heart Block (Cardiac disorders) | 2 (2)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1)
Heart Valve Incompetence (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2)
Mitral Valve Disease (Cardiac disorders) | 2 (2)
Mitral Valve incompetence (Cardiac disorders) | 2 (2)
Mitral Valve stenosis (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 9 (9)
Nodal Rhythm (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Right ventricular failure (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 29 (29)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular asystole (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 4 (4)
Ventricular dysfunction (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 4 (4)
Left ventricular outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Colonic pseudo obstruction (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 15 (15)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 6 (6)
Intestinal perforation (Gastrointestinal disorders) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 14 (14)
Gait disturbance (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 6 (6)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 3 (3)
Porcelain gallbladder (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5)
Cellulitis (Infections and infestations) | 4 (4)
Central line infection (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 7 (7)
Diverticlitis (Infections and infestations) | 4 (4)
Empyema (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 5 (5)
Enterococcal infection (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Graft infection (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 36 (36)
Wound infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 18 (18)
Septic shock (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural thoracic complication (Injury, poisoning and procedural complications) | 4 (4)
Traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemotoma (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 4 (4)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Decreased mobility (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osterarthritis (Musculoskeletal and connective tissue disorders) | 8 (8)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anoxic encephalopothy (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Coratid artery stenosis (Nervous system disorders) | 2 (2)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 13 (13)
Dementia (Nervous system disorders) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Facial paresis (Nervous system disorders) | 1 (1)
Hemianopia homonymous (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Anorexia nervosa (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 32 (32)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 40 (40)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 65 (65)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac pacemaker revision (Surgical and medical procedures) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 3 (3)
Mitral valve replacement (Surgical and medical procedures) | 1 (1)
Vertebroplasty (Surgical and medical procedures) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2)
Arterial insufficiency (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 19 (19)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 13 (13)
Peripheral vascular disorder (Vascular disorders) | 3 (3)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=365)
Aenemia (Blood and lymphatic system disorders) | 22 (22)
Hypotension (Vascular disorders) | 27 (30)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 59 (59)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 31 (31)
Renal Failure (Renal and urinary disorders) | 48 (48)
Pneumonia (Infections and infestations) | 22 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 (28)
Urinary Tract Infection (Renal and urinary disorders) | 38 (42)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT01694563/Prot_SAP_000.pdf